CLINICAL TRIAL: NCT05585099
Title: Effects of Retro Walking Exercise Using Lower Body Positive Pressure on Knee Pain and Physical Function in People With Knee Osteoarthritis
Brief Title: Effects of Lower Body Positive Pressure in People With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Sattam Almutairi, Assistant professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-07-07
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will walk in retro walking exercise on lower body positive pressure treadmill.
  Interventions: Other: Exercise
- Control (Other): Participants will walk in forward walking exercise on lower body positive pressure treadmill.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will stand on lower body positive pressure treadmill and participate in walking exercise.
  Other Names: Walking exercise

SUMMARY:
The goal of this clinical trial is to compare effects of retro walking exercise versus forward walking using lower body positive pressure on knee pain, physical function, and quadriceps muscle strength in people with mild to moderate knee OA. The secondary aim is to compare effects of retro walking exercise versus forward walking using lower body positive pressure on mobility function, balance, and self-reported health outcomes in people with mild to moderate knee OA. The main questions it aims to answer are:

* Does retro walking exercise improve knee pain, physical function and Quadriceps muscle strength compared to forward walking exercise using lower body positive pressure in people with mild to moderate knee osteoarthritis?
* Does retro walking exercise improve Mobility function, balance, and self-reported health outcomes compared to forward walking exercise using lower body positive pressure in people with mild to moderate knee osteoarthritis?

Participants will walk (retro versus forward) on a lower body positive pressure treadmill.

If there is a comparison group: Researchers will compare [retro walking compares to forward walking] to see if [improve in knee pain, physical function, and quadriceps muscles strength]

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate knee osteoarthritis
* Edge bigger or equal 40 years
* Knee pain reported by participants in the past 30 days
* One or both knees osteoarthritis graded with Kellgren & Lawrence grade 1 - 3

Exclusion Criteria:

* If they didn't meet the inclusion criteria
* History of hip, knee or ankle injury or surgery within the last year
* Kellgren & Lawrence grade > 3 of severe knee OA
* Diagnosed with rheumatoid arthritis
* History of knee injection with any medicine that reduce pain within the last year
* History of other medical condition that would disturb normal walking function
* Receive physical therapy in the last three months
* Pregnant
* Other conditions that are Contra indication to lower body positive pressure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | Change from baseline pain at 6 weeks
  The NPRS is an 11-point scale with "0" representing "no pain" and "10" representing "most imaginable pain" used to assess pain intensity.
Knee injury and osteoarthritis outcome score (KOOS) | Change from baseline pain, symptoms, and level of disability at 6 weeks.
  The KOOS is a self-reported, knee-specific questionnaire that is aimed to measure knee pain, symptoms, and level of disability during the last week.
Thigh muscle strength test | Change from baseline thigh muscle strength at 6 weeks.
  A Biodex isokinetic dynamometer (Model 4Pro) connected to a computer will be used to assess bilateral knee's flexor and extensor isometric muscle strength.

SECONDARY OUTCOMES:
Five times sit to stand test | Change from baseline balance at 6 weeks.
  The FTSST is used to assess lower extremity strength and balance and is an indicator of postural control.
3-M Backward Walk Test | Change from baseline backward walking at six weeks.
  Patients will be instructed to walk backwards when the assessor says "go" and stop when the participant pass the end line colored tape. The participant will be allowed to look back.
Timed up and go test | Change from baseline Functional mobility at six weeks.
  The TUG assesses functional mobility by assessing an individual's ability to stand up, walk 3 meters at a comfortable pace, turn 180 degrees, walk back 3 meters, and sit down
4 square step test | Change from baseline dynamic balance and coordination at six weeks
  The test is designed to assess dynamic balance and coordination.
Functional reach test | Change from baseline static balance at six weeks
  FRT used to assess participant's stability and balance by measuring the maximum distance participant can reach forward while standing in fixed position.
10-Meter Walk Test | Change from baseline walking speed at six weeks
  The 10-MWT evaluates walking speed over a short duration with or without an assistive device.
6 minute walk test | Change from baseline aerobic capacity and endurance at six week
  6MWT assesses the distance walked over 6 minutes as a test of aerobic capacity and endurance.
Medical Outcomes Study Short Form 12 (SF-12) | Change from baseline quality of life at six weeks
  It is a health survey that evaluates health related quality of life in a clinical practice and research purpose
Patient Health Questionnaire -9 | Change from baseline depression at six week
  PHQ-9 is an instrument to evaluate depression symptoms among different populations.
Rapid Assessment of Physical Activity | Change from baseline physical activity at six week
  RAPA is a 9-items, self-reported questionnaire measures the levels of physical activity of adult older than 50 years.

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Qassim university medical city, Buraidah, Almuledia
  - Medical City in Qassim University, Buraidah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almutairi SM, Almutairi MK, Alotaibi MM, Alshehri M, Alenazi AM. Effects of backward walking exercise using lower body positive pressure treadmill on knee symptoms and physical function in individuals with knee osteoarthritis: a protocol for RCT. J Orthop Surg Res. 2023 Apr 1;18(1):264. doi: 10.1186/s13018-023-03711-x. PMID 37005596